CLINICAL TRIAL: NCT04929600
Title: Prospective Comparison of Angiotensin Receptor Neprilysin Inhibitor (ARNI) With Amlodipine on Ventricular Remodeling in Hypertension and Left Ventricular Hypertrophy.
Brief Title: Sacubitril/Valsartan Versus Amlodipine in Hypertension and Left Ventricular Hypertrophy.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PARASTRAIN
Record Dates: First submitted 2021-06-15; First posted 2021-06-18 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Hypertension; Left Ventricular Hypertrophy
Keywords: sacubitril/valsartan; amlodipine; blood pressure; global longitudinal strain
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — sacubitril and valsartan sodium hydrate drug combination; Amlodipine

STUDY DESIGN:
Intervention Model Description: After screening and run-in period, eligible patients will be randomly assigned into ARNI group (sacubitril/valsartan 200-400mg QD) or amlodipine group (amlodipine 5-10mg QD).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients in ARNI group will take sacubitril/valsartan + matching placebo of amlodipine; Patients in amlodipine group will take amlodipine + matching placebo of sacubitril/valsartan. Any markers that can identify placebo or active drugs will be removed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): One pill of sacubitril/valsartan (200mg tablet) + one pill of matching placebo of amlodipine daily. If possible, dosage titration should be conducted.
  Interventions: Drug: sacubitril/valsartan
- Comparator (Active Comparator): One pill of amlodipine (5mg tablet) + one pill of matching placebo of sacubitril/valsartan daily. If possible, dosage titration should be conducted.
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: sacubitril/valsartan — Sacubitril/valsartan oral tablets (200mg) one pill a day + matching placebo of amlodipine one pill a day.
  Arms: Experimental
Drug: Amlodipine — Amlodipine oral tablets (5mg) one pill a day + matching placebo of sacubitril/valsartan one pill a day.
  Arms: Comparator

SUMMARY:
1. Study name: Prospective Comparison of Angiotensin receptor neprilysin inhibitor (ARNI) with Amlodipine on ventricular remodeling in hypertension and left ventricular hypertrophy.
2. Medicine: sacubitril/valsartan (ARNI, 200mg tablet) and the matching placebo; amlodipine (5mg tablet) and the matching placebo.
3. Rationale: according to the results of previous clinical studies, ARNI has obvious advantages in improving cardiac remodeling and reducing blood pressure. However, there is no evidence to demonstrate the efficacy of ARNI in reducing blood pressure and improving ventricular remodeling in hypertension patients with left ventricular hypertrophy (LVH) compared with calcium channel blockers.
4. Objective: to demonstrate the superior efficacy of ARNI on improvement of LVH and blood pressure control compared with amlodipine in hypertension patients with LVH.
5. Study design: This study This is a 24-week prospective, randomized, active-controlled, double-blind, multi-center study, with two equally sized treatment groups: sacubitril/valsartan (200mg tablet); amlodipine (5mg tablet).
6. Study population: men or women aged over 18 years; Untreated patients or patients with taking single antihypertensive drugs; Essential mild to moderate hypertension; Echocardiographic diagnosis of LVH.
7. Randomization and treatment: Eligible patients will be randomly divided into 2 groups, taking one pill of sacubitril/valsartan (200mg tablet) + one pill of matching placebo of amlodipine daily, or one pill of amlodipine (5 mg/tablet) + one pill of matching placebo of sacubitril/valsartan daily.
8. Follow up: after meeting the inclusion criteria, there will be 2-week placebo run-in. Then patients will be randomly assigned into ARNI group and amlodipine group. There will be 5 visiting points in the treatment period, which will be the 4th week, 8th week, 12th week, 18th week and 24th week.
9. Sample size: 120 patients in total.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in April 2021, recruitment will start. Patients enrollment and follow-up will be performed between June 2021 to June 2022.

DETAILED DESCRIPTION:
1. Study name: Prospective Comparison of Angiotensin receptor neprilysin inhibitor (ARNI) with Amlodipine on ventricular remodeling in hypertension and left ventricular hypertrophy.
2. Medicine: sacubitril/valsartan (ARNI, 200mg tablet) and the matching placebo; amlodipine (5mg tablet) and the matching placebo.
3. Rationale: according to the results of previous clinical studies, ARNI has obvious advantages in improving cardiac remodeling and reducing blood pressure. However, there is no evidence to demonstrate the efficacy of ARNI in reducing blood pressure and improving ventricular remodeling in hypertension patients with left ventricular hypertrophy (LVH) compared with calcium channel blockers.
4. Objective: to demonstrate the superior efficacy of ARNI on improvement of LVH and blood pressure control compared with amlodipine in hypertension patients with LVH.
5. Study design: This study This is a 24-week prospective, randomized, active-controlled, double-blind, multi-center study, with two equally sized treatment groups: sacubitril/valsartan (200mg tablet); amlodipine (5mg tablet).
6. Study population: men or women aged over 18 years will be screened for hypertension and LVH. Eligible patients should be untreated patients or patients with taking single antihypertensive drugs with essential mild to moderate hypertension (clinic systolic blood pressure ≥ 140 and < 180mmHg), and echocardiographic diagnosis of LVH (LVMI: male≥115g/m2, female≥ 95g/m2). Patients should have abilities to understand the study requirements and provide informed consent.
7. Randomization and treatment: After screening period and run-in period by centers, eligible patients will be randomly divided into 2 groups, taking one pill of sacubitril/valsartan (200mg tablet) + one pill of matching placebo of amlodipine daily, or one pill of amlodipine (5 mg/tablet) + one pill of matching placebo of sacubitril/valsartan daily. At the 12th week of treatment, if systolic blood pressure ≥ 120 mmHg or diastolic blood pressure ≥ 80 mmHg and no safety problems, dosage titration (sacubitril/valsartan 200mg QD to 400mg QD, amlodipine 5mg QD to 10mg QD) should be conducted.
8. Follow up: after meeting the inclusion criteria, there will be 2-week placebo run-in. Clinic blood pressure, ambulatory blood pressure, echocardiography, NT proBNP, myocardial fibrosis index, concomitant medication records and adverse event records will be collected at randomization/the end of run-in period. Then patients will be randomly assigned into ARNI group and amlodipine group. The treatment will be observed for 24 weeks. There will be 5 visiting points in the treatment period, which will be the 4th week, 8th week, 12th week, 18th week and 24th week. Global longitudinal strain (GLS) was detected at randomization, the 12th week and 24th week.
9. Sample size: At least 60 eligible patients should be enrolled in each group, and a total of 120 patients should be enrolled in total.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in April 2021, recruitment will start. Patients enrollment and follow-up will be performed between June 2021 to June 2022.
11. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18;
* Essential mild to moderate hypertension (office systolic blood pressure (SBP) ≥ 140 and < 180mmHg in untreated patients or patients with taking single antihypertensive drugs (not including single-pill combination))；
* Echocardiographic diagnosis of LVH，LVMI: male≥115g/m2, female≥ 95g/m2;
* Ability to understand the study requirements and provide informed consent.

Exclusion Criteria:

* Hypersensitivity history to any study drug or similar drug (ARB, ACEI, neprilysin inhibitor；
* Severe renal insufficiency (eGFR < 30 mL/min/1.73m2);
* Hyperkalemia (serum potassium > 5mmol/L);
* Active liver disease or hepatic insufficiency (AST or ALT > 3 times upper limit of normal);
* History of malignancy over the past 5 years;
* Severe disease patients with life expectancy of < 1 year;
* Previous or current diagnosis of heart failure;
* Stroke or myocardial infarction within 6 months;
* Previous or current atrial fibrillation, frequent ventricular premature beats, supraventricular tachycardia;
* Patients who are receiving other study drugs or study medical devices;
* Pregnant or lactating women;
* Other circumstances that patients are not appropriate for the study upon the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-28 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in LVGLS after 24 weeks | Baseline and 24 weeks
  Change in left ventricular global longitudinal strain (LVGLS) after 24-week treatments. At baseline and 24-week follow-up, all patients will undergo standard transthoracic echocardiography performed in the sinus rhythm using the Vivid E9 and E95 Echo-system (General Electric Medical Health, Milwaukee, Wisconsin, USA) equipped with a M5S transducer. LVGLS will be obtained from two-, three-, and four-chamber apical views, and LVGLS analysis will be performed using an offline software (EchoPac, Version 113; General Electric Medical Health).

SECONDARY OUTCOMES:
Change in LVGLS after 12 weeks | Baseline and 12 weeks
  Change in left ventricular global longitudinal strain (LVGLS) after 12-week treatments. At baseline and 12-week follow-up, all patients will undergo standard transthoracic echocardiography performed in the sinus rhythm using the Vivid E9 and E95 Echo-system (General Electric Medical Health, Milwaukee, Wisconsin, USA) equipped with a M5S transducer. LVGLS will be obtained from two-, three-, and four-chamber apical views, and LVGLS analysis will be performed using an offline software (EchoPac, Version 113; General Electric Medical Health).
Changes in LVMI after 24 weeks | Baseline and 24 weeks
  At baseline and 24-week follow-up, all patients will undergo standard transthoracic echocardiography, Images of parasternal long axis view will be recorded to measure left ventricular end-diastole diameter (LVEDD), interventricular septal (IVS) and left ventricular posterior wall thickness (LVPW), and left ventricular mass will be calculated using the formula: 0.8*{1.04*[(LVEDD+IVS+LVPW)^3-LVEDD^3]}+0.6, and indexed by body surface area (BSA) as left ventricular mass index (LVMI).
Changes in LVMI after 12 weeks | Baseline and 12 weeks
  At baseline and 12-week follow-up, all patients will undergo standard transthoracic echocardiography, Images of parasternal long axis view will be recorded to measure left ventricular end-diastole diameter (LVEDD), interventricular septal (IVS) and left ventricular posterior wall thickness (LVPW), and left ventricular mass will be calculated using the formula: 0.8*{1.04*[(LVEDD+IVS+LVPW)^3-LVEDD^3]}+0.6, and indexed by body surface area (BSA) as left ventricular mass index (LVMI).
Blood pressure after 24 weeks | Baseline and 24 weeks
  Changes in clinic blood pressure, ambulatory blood pressureover 24 hours, daytime and nighttime after 24-week treatments.
Blood pressure after 12 weeks | Baseline and 12 weeks
  Changes in clinic blood pressure, ambulatory blood pressureover 24 hours, daytime and nighttime after 12-week treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China